CLINICAL TRIAL: NCT05412212
Title: A Brief Educational Video for Patients Prescribed Latent Tuberculosis Treatment: A Randomized Trial in an Integrated Healthcare Organization in the United States
Brief Title: Brief Educational Video for Patients Prescribed LTBI Treatment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 12324
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Latent Tuberculosis
Keywords: adherence; digital health intervention
MeSH Terms: conditions — Latent Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LTBI video intervention (Experimental): Patients randomized to the intervention group will be sent an invitation with a link to watch a brief (~3 minute video) about the importance of taking and completing LTBI treatment.
  Interventions: Other: LTBI video intervention
- Standard care (No Intervention): Patients who are randomized to receive standard of care will not receive any messages or have any contact with the research team.

INTERVENTIONS:
Other: LTBI video intervention — 3-minute educational video about latent tuberculosis and importance of taking and completing treatment
  Arms: LTBI video intervention

SUMMARY:
Many patients who are prescribed treatment for latent tuberculosis (LTBI) do not complete treatment. Effective interventions that are low-cost and feasible for large-scale implementation are needed to support efforts to eliminate TB. The investigators hypothesize that a 3-minute educational LTBI video intervention will improve treatment completion compared to standard care (no intervention).

A randomized trial will be conducted at Kaiser Permanente Southern California, including adults who are prescribed treatment for LTBI, identified using an electronic health record algorithm. At the time of treatment prescription, patients will be randomized to receive the LTBI video intervention or standard care at a ratio of 2 to 1. Those in the intervention group will be sent a secure text message or e-mail with a link to the video. Individuals who watch the LTBI video will be invited to respond to 4 short questions about their perceptions of the video accessibility and content.

The primary outcome is LTBI treatment completion (dispensation of the required number of doses) in the year following prescription order. Secondary outcomes are LTBI treatment initiation (at least one dispensation) in the year following prescription order; initiation and completion within the year following prescription order stratified by LTBI treatment regimen (if feasible); the proportion of individuals randomized to the intervention group who watched the LTBI video; and the perceptions of those who watched the video.

The primary analysis will be based on intention-to-treat. Characteristics of individuals in the intervention and standard care groups will be described, and rates of LTBI treatment completion will be calculated. To assess the effect of the intervention, Poisson regression with robust standard errors will be used to estimate unadjusted and adjusted rate ratios and 95% confidence intervals. Per-protocol analyses will also be conducted, comparing those in the intervention group who watched the LTBI video to those in the standard care group. Similar methods will be used for secondary analyses.

Assuming the completion rate in the standard care group is 0.5 (based on recent KPSC data), approximately 918 patients will be needed to achieve 80% power with type one error 0.05 to detect an intervention effect of 0.10 in the completion rate between groups. This sample size will be feasible to achieve over the 1 year trial duration.

DETAILED DESCRIPTION:
Please see the full protocol for details of the study.

ELIGIBILITY:
Inclusion criteria:

* Active KSPC member
* Age ≥18 years
* Receipt of an LTBI treatment prescription order (medication ID codes listed below)

  * Isoniazid: 12199066, 1214000023, 1216000272, 12022505, 12035328, 12035329, 12035330, 12035331, 12035332, 12035333, 12035334, 12035335, 12035336, 12035337, 12015833, 12032230, 12035338, 12035339, 12035340, 12035341, 12035342, 12035343, 12035344, 12035345, 12024985, 12035346, 12181973
  * Rifampin: 12199042, 121103412, 1214000029, 1214000030, 1214000340, 1214000565, 1215200240, 1206096, 12017860, 1209060, 12011205, 12015920, 190716, 1902899, 190207268, 190210700, 12189972, 12189977, 12189987
  * Isoniazid (see codes above) + Rifampin (see codes above), also: 12032976, 12199041, 12029484, 12189973, 12168828
  * Isoniazid (see codes above) + Rifapentine (121100982, 1206442, 12025808, 12188784, 12189978)
* LTBI ICD-10 diagnosis code prior to prescription order: R76.11, R76.12, Z22.7

Exclusion Criteria:

• Active TB ICD-10 diagnosis code prior to prescription order: A15, A17, A18, A19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1898 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2024-12-29 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment completion | 1 year after treatment prescription
  Proportion of patients prescribed LTBI treatment who complete the treatment within one year of treatment prescription

SECONDARY OUTCOMES:
Treatment initiation | 1 year after treatment prescription
  Proportion of patients prescribed LTBI treatment who initiate the treatment within one year of treatment prescription
Treatment initiation by treatment regimen | 1 year after treatment prescription
  Proportion of patients prescribed LTBI treatment who initiate the treatment within one year of treatment prescription, by treatment regimen (if feasible)
Treatment completion by treatment regimen | 1 year after treatment prescription
  Proportion of patients prescribed LTBI treatment who complete the treatment within one year of treatment prescription, by treatment regimen (if feasible)
Video Watch Completion | 1 year after treatment prescription
  Proportion of patients randomized to the LTBI video who watch the full video
Video Accessibility | 1 year after treatment prescription
  Proportion of patients who watch the video who report no difficulties watching the video
Understanding of Treatment Importance | 1 year after treatment prescription
  Proportion of patients who watch the video who report understanding the importance of completing LTBI treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente Southern California Department of Research and Evaluation, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/12/NCT05412212/Prot_001.pdf